CLINICAL TRIAL: NCT01947907
Title: A Multicenter, Phase 2, Randomized, Open Label, Active-controlled, Parallel-group Study Investigating the Safety, Tolerability, and Efficacy of Different Dose Levels of ACP-001 Administered Once Weekly Versus Standard Daily rhGH Replacement Therapy in Pre-pubertal Children With Growth Hormone Deficiency (GHD)
Brief Title: Safety, PK/PD (Pharmacokinetics/Pharmacodynamics) and Efficacy of ACP-001 Weekly Versus Daily hGH in Children With Growth Hormone Deficiency (GHD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ascendis Pharma A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACP-001_CT-004
Record Dates: First submitted 2013-06-03; First posted 2013-09-23 (Estimated); Results first posted 2017-01-19 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2016-11

CONDITIONS: Growth Hormone Deficiency (GHD)
Keywords: Human Growth Hormone; rhGH; hGH; GHD
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ACP-001, dose-level 1 (Experimental): Once weekly subcutaneous injection of ACP-001
  Interventions: Drug: ACP-001
- ACP-001, dose-level 2 (Experimental): Once weekly subcutaneous injection of ACP-001
  Interventions: Drug: ACP-001
- ACP-001, dose-level 3 (Experimental): Once weekly subcutaneous injection of ACP-001
  Interventions: Drug: ACP-001
- Human Growth Hormone (Active Comparator): Once daily subcutaneous injection of human Growth Hormone (rhGH)
  Interventions: Drug: Human Growth Hormone

INTERVENTIONS:
Drug: ACP-001 — Once weekly subcutaneous injection
  Arms: ACP-001, dose-level 1; ACP-001, dose-level 2; ACP-001, dose-level 3
Drug: Human Growth Hormone — Once daily subcutaneous injection of human Growth Hormone
  Other Names: Somatropin
  Arms: Human Growth Hormone

SUMMARY:
A six month study of ACP-001, a long-acting growth hormone product, versus standard human growth hormone therapy. ACP-001 will be given once-a-week, standard human growth hormone (hGH) will be given on a daily basis. The primary aim is to demonstrate safety, pharmacokinetics and pharmacodynamics over a period of six months. A secondary objective is the comparison of height velocity (HV) of the ACP-001 treated groups to the daily hGH treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Prepubertal children, Tanner stage 1
* Diagnosis of GHD, confirmed by two stimulation tests
* Bone age not greater than chronological age
* Impaired height and height velocity
* BMI within +/- 2 SD (standard deviations)
* Baseline IGF-1 (insulin-like growth factor)
* Normal fundoscopy
* Stable hormonal replacement therapy (other than hGH)
* Written Informed Consent

Exclusion Criteria:

* Prior exposure to rhGH or IGF-I
* Past or present intracranial tumor; history or presence of malignant disease
* Small for gestational age (SGA)
* Malnutrition
* Psychosocial dwarfism
* Coeliac disease
* Anti-hGH antibodies
* Diabetes mellitus
* Chromosomal abnormalities (e.g. Turner syndrome, SHOX)
* Closed epiphyses
* Known or suspected HIV infection

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2013-07; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Chatelain, Prof, MD, Principal Investigator — University of Lyon; Michael Beckert, MD, Study Director — Ascendis Pharma A/S
Locations (36):
- 2nd Children City Clinic, Minsk, Belarus
- University Multiprofile Hospital for Active Treatment (UMHAT) "Sv. Marina", Varna, Bulgaria
- Masaryk´s Hospital, Ústí nad Labem, Czechia
- Egypt (4):
  - El Shatby University Hospital, Alexandria
  - Ain Shams University Hospital, Cairo
  - Cairo University Hospital, Cairo
  - El Mansoura University Hospital, El Mansoura
- France (3):
  - Hôpital des enfants Pellegrin, Bordeaux
  - Hôpital Jeanne de Flandre, Lille
  - Hôpital Femme-Mère-Enfant, Lyon
- Germany (2):
  - University Hospital Leipzig, Leipzig
  - University Children's Hospital Magdeburg, Magdeburg
- Children's Hospital of Athens "P. A. Kyriakou", Athens, Greece
- Hungary (4):
  - Buda Children's Hospital, Budapest
  - Heim Pal Children's Hospital, Budapest
  - University of Pecs, Pécs
  - University of Szeged, Szeged
- Poland (4):
  - University Medical Hospital, Katowice
  - Medical University of Lublin, Lublin
  - Regional Hospital N°2 Rzeszow, Rzeszów
  - Children's Memorial Health Institute Warsaw, Warsaw
- Romania (3):
  - Emergency Clinical Hospital Cluj-Napoca, Cluj-Napoca
  - St. Spiridon County Clinic Emergency Hospital, Iași
  - Louis Turcanu Emergency Hospital for Children Timisoara, Timișoara
- Russia (4):
  - Federal State Budgetary Institution, Moscow
  - St. Petersburg State Pediatric Medical Academy, Saint Petersburg
  - Samara State Medical University, Samara
  - Bashkir State Medical University, Ufa
- Children's University Hospital, Ljubljana, Slovenia
- Turkey (Türkiye) (2):
  - Ankara University School of Medicine, Ankara
  - Ege Üniversity, Izmir
- Ukraine (5):
  - Donetsk Regional Children Clinical Hospital, Donetsk
  - Kharkiv National Medical University, Kharkiv
  - Institute of Endocrinology and Metabolism, Kiev
  - Ukrainian Children Specialized Clinical Hospital, Kiev
  - Odessa National Medical University, Odesa

REFERENCES:
- [Derived] Chatelain P, Malievskiy O, Radziuk K, Senatorova G, Abdou MO, Vlachopapadopoulou E, Skorodok Y, Peterkova V, Leff JA, Beckert M; TransCon GH Working Group. A Randomized Phase 2 Study of Long-Acting TransCon GH vs Daily GH in Childhood GH Deficiency. J Clin Endocrinol Metab. 2017 May 1;102(5):1673-1682. doi: 10.1210/jc.2016-3776. PMID 28201598

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ACP-001, Dose-level 1 | ACP-001, Dose-level 2 | ACP-001, Dose-level 3 | Human Growth Hormone
Started | 12 | 14 | 14 | 13
Completed | 12 | 14 | 14 | 13
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACP-001, Dose-level 1 | ACP-001, Dose-level 2 | ACP-001, Dose-level 3 | Human Growth Hormone | Total
Number analyzed (Participants) | 12 | 14 | 14 | 13 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 14 | 14 | 13 | 53
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.98 (2.889) | 8.24 (2.13) | 7.32 (2.784) | 7.53 (2.483) | 7.77 (2.57)
Gender [Count of Participants; unit: Participants]
  Female | 3 | 4 | 5 | 3 | 15
  Male | 9 | 10 | 9 | 10 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 12 | 14 | 14 | 13 | 53
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Russian Federation | 4 | 4 | 7 | 6 | 21
  Romania | 1 | 0 | 0 | 1 | 2
  Hungary | 0 | 0 | 1 | 0 | 1
  Egypt | 2 | 4 | 0 | 1 | 7
  Ukraine | 1 | 4 | 1 | 1 | 7
  Belarus | 2 | 2 | 2 | 1 | 7
  Greece | 1 | 0 | 2 | 0 | 3
  Turkey | 1 | 0 | 0 | 2 | 3
  Poland | 0 | 0 | 1 | 0 | 1
  Bulgaria | 0 | 0 | 0 | 1 | 1
Baseline IGF-1 SDS (standard deviation score) [Mean (Standard Deviation); unit: Standard Deviation Score] | -2.034 (0.7429) | -2.017 (0.7713) | -2.19 (0.7169) | -2.502 (0.896) | -2.19 (0.782)
Baseline Height SDS [Mean (Standard Deviation); unit: Standard Deviation Score] | -3.05 (1.127) | -2.75 (0.383) | -3.17 (1.04) | -3.27 (1.077) | -3.06 (0.905)
Screening Peak GH Values [Mean (Standard Deviation); unit: ng/mL] | 5.09 (3.169) | 5.16 (2.598) | 4.44 (2.770) | 5.15 (3.068) | 4.95 (2.829)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Anti-hGH Binding Antibody Formation
Description: Number of subjects with positive results for anti-hGH binding antibodies at two consecutive post-dose visits
Time Frame: Visit 2 - Visit 5
Population: Safety analysis set includes all patients who receive at least one dose of planned study medication
Measure: Number; unit: participants
Arm/Group | ACP-001, Dose-level 1 | ACP-001, Dose-level 2 | ACP-001, Dose-level 3 | Human Growth Hormone
Number analyzed (Participants) | 12 | 14 | 14 | 13
participants | 1 | 0 | 0 | 0

2. Primary Outcome: Incidence of Anti-hGH Neutralizing Antibody Formation
Description: Number of subjects with positive results for anti-hGH neutralizing antibodies at two consecutive post-dose visits
Time Frame: Visit 2 - Visit 5
Measure: Number; unit: participants
Arm/Group | ACP-001, Dose-level 1 | ACP-001, Dose-level 2 | ACP-001, Dose-level 3 | Human Growth Hormone
Number analyzed (Participants) | 12 | 14 | 14 | 13
participants | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Subjects Reporting Local Tolerability Events (Assessed by the Patient and Investigator)
Description: Assessment of local tolerability was performed by examining injection sites (by the investigator during study visits) and on the basis of anamnestic data and records in the Patient Diary. Assessments included pain, redness, bruising, swelling, and itching. Every subject was counted only once within each symptom category.
Time Frame: Start of study treatment through Visit 5 (Week 27)
Measure: Number; unit: Number of subjects with any symptom
Arm/Group | ACP-001, Dose-level 1 | ACP-001, Dose-level 2 | ACP-001, Dose-level 3 | Human Growth Hormone
Number analyzed (Participants) | 12 | 14 | 14 | 13
Number of subjects with any symptom | 7 | 6 | 6 | 6

4. Primary Outcome: Cmax of hGH
Description: As part of the following endpoint:
  PK profile of serum hGH from ACP-001 treated patients compared between ACP-001 dose groups and to the pharmacokinetic (PK) profile of hGH from the daily rhGH groups during visit 1 and 3.
  Uncorrected Cmax (maximum value of concentration) values at Visit 3 (Week 13)
Time Frame: 0 hours to 168 hours at Visit 3 (Week 13)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ACP-001, Dose-level 1 | ACP-001, Dose-level 2 | ACP-001, Dose-level 3 | Human Growth Hormone
Number analyzed (Participants) | 12 | 14 | 14 | 13
ng/mL | 12.558 (8.678) | 13.418 (9.428) | 31.8 (17.499) | 16.612 (12.777)

5. Primary Outcome: AUC0-168h of hGH
Description: As part of the following endpoint:
  PK profile of serum hGH from ACP-001 treated patients compared between ACP-001 dose groups and to the PK profile of hGH from the daily rhGH group during Visit 1 and Visit 3
  Uncorrected AUC0-168h (area under the curve from 0h to 168h) values at Visit 3 (Week 13)
Time Frame: 0 hours to 168 hours at Visit 3 (Week 13)
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | ACP-001, Dose-level 1 | ACP-001, Dose-level 2 | ACP-001, Dose-level 3 | Human Growth Hormone
Number analyzed (Participants) | 12 | 14 | 14 | 13
h*ng/mL | 696.34 (410.096) | 787.41 (483.169) | 2167.43 (1064.729) | 556.88 (412.618)

6. Primary Outcome: E-Trough of IGF-1
Description: As part of the following endpoint:
  PD profile of serum IGF-1 during Visit 1 and Visit 3 compared between the ACP-001 dose groups and to the daily rhGH group
  Uncorrected E-Trough (the pre-dose efficacy response) values at Week 13
Time Frame: 0 hours to 168 hours at Visit 3 (Week 13)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ACP-001, Dose-level 1 | ACP-001, Dose-level 2 | ACP-001, Dose-level 3
Number analyzed (Participants) | 12 | 14 | 14
ng/mL | 97.17 (50.53) | 156 (76.235) | 167.83 (74.01)

7. Primary Outcome: Emax of IGF-1
Description: As part of the following endpoint:
  PD profile of serum IGF-1 during V1 and V3 compared between the ACP-001 dose groups and to the daily rhGH group
Time Frame: 0 hours to 168 hours at Visit 3 (Week 13)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ACP-001, Dose-level 1 | ACP-001, Dose-level 2 | ACP-001, Dose-level 3
Number analyzed (Participants) | 12 | 14 | 14
ng/mL | 209.5 (120.189) | 276 (126.632) | 289.92 (129.469)

8. Primary Outcome: AUEC0-168h of IGF-1
Description: As part of the following endpoint:
  PD profile of serum IGF-1 during V1 and V3 compared between the ACP-001 dose groups and to the rhGH group.
  Uncorrected AUEC0-168 (area under the efficacy curve from 0h-168h) values at Week 13
Time Frame: 0 hours to 168 hours at Visit 3 (Week 13)
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | ACP-001, Dose-level 1 | ACP-001, Dose-level 2 | ACP-001, Dose-level 3
Number analyzed (Participants) | 12 | 14 | 14
h*ng/mL | 28526.19 (15756.44) | 35591.94 (17068.59) | 36066.01 (17379.44)

9. Secondary Outcome: Annualized Height Velocity
Description: Annualized HV during treatment with ACP-001 or daily rhGH at the end of 6 months, for each ACP-001 dose group and for the daily rhGH dose group
Time Frame: Baseline to 6 months (Visit 5)
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | ACP-001, Dose-level 1 | ACP-001, Dose-level 2 | ACP-001, Dose-level 3 | Human Growth Hormone
Number analyzed (Participants) | 12 | 14 | 14 | 13
cm/year | 11.93 (4.066) | 12.89 (3.464) | 13.85 (4.009) | 11.64 (3.592)

ADVERSE EVENTS:
Time Frame: From start of the study treatment and continues until the end of the patient's participation in the study (until 4 weeks after stop of patient's study participation for serious adverse events)
Arm/Group | ACP-001, Dose-level 1 | ACP-001, Dose-level 2 | ACP-001, Dose-level 3 | Human Growth Hormone
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/14 | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 7/12 | 6/14 | 8/14 | 8/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACP-001, Dose-level 1 (N=12) | ACP-001, Dose-level 2 (N=14) | ACP-001, Dose-level 3 (N=14) | Human Growth Hormone (N=13)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACP-001, Dose-level 1 (N=12) | ACP-001, Dose-level 2 (N=14) | ACP-001, Dose-level 3 (N=14) | Human Growth Hormone (N=13)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperthermia (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Heat exhaustion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Open wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood triglycerides (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thalassemia beta (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Iron deficiency anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Strabismus (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal pruritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Secondary hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tonsilitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth abcess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No